CLINICAL TRIAL: NCT04092348
Title: Value of FoxO3a and PU.1 Expression in Pediatric Acute Lymphoblastic Leukemia
Brief Title: FoxO3a and PU.1 in Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MRA Youb, principal investigator, Assiut University
Other Study IDs: madonna
Record Dates: First submitted 2019-09-14; First posted 2019-09-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: children aged 2-17 years and diagnosed as new cases of acute lymphoblastic leukemia
  Interventions: Other: complete blood count
- control group: healthy age- and sex-matched children without ahistory of any malignancies
  Interventions: Other: complete blood count

INTERVENTIONS:
Other: complete blood count — 1. total RNA is isolated from fresh blood samples
  2. RNA is converted into complementary DNA c.DNA
  3. cDNA is then analysed by quantitatine Real Time PCR(qRT-PCR) to evaluate the relative expression levels of FoxO3a, PU.1 genes and TATA-binding protein (TBP) ,as an endogenous control gene.
  Other Names: bone marrow aspirate

SUMMARY:
Acute Lymphoblastic Leukemia (ALL) is one of the four major types of leukemia which is common in both children and adolescents; however, it is the most common pediatric malignancy diagnosed in children younger than 20 years .The disease pathogenesis results from blockade at any stages of normal lymphoid differentiation with uncontrolled proliferation of lymphoid cells. According to the World Health Organization (WHO) definition, ALL is categorized in B-Lymphoblastic Leukemia (B-ALL) And T-Lymphoblastic Leukemia (T-ALL), originated from B- and T-Lineage lymphoid precursor cells, respectively.

DETAILED DESCRIPTION:
Proto-oncogenes and tumor suppressor genes are the most important genes involved in leukemogenesis , which their alterations disrupt normal regulatory processes such as self-renewal, proliferation, differentiation and apoptosis in target cells. Among those genes FoxO3a gene and PU.1 gene.

FoxO(Fork head box ,class O) transcription factors function as a tumor suppressor gene and are important for stem cell maintenance.They are key regulators of the cellular differentiation, growth, survival, cell cycle, metabolism, and cellular stress. There are four members of the foxO transcription factors in humans : foxO1, foxO3a, foxO4, foxO6 .FoxO3a is expressed in various tissues including B - and T-lymphoid cells. Over expression of FoxO3a in B and T cell lines induces cell cycle arrest in G1 phase , so it inhibits cell proliferation . FoxO3a is an important target of PI3K/AKT signaling pathway,which is hyperactivated in various types of cancers .Hyperactivation of this pathway in leukemia leads to inactivation of foxO3a in leukemic cells and enhances tumor growth .

PU .1(Purine-rich box 1) is a member of the E26 transformation-specific (ETS) Family . Normal hematopoiesis is securely controlled by asmall number of lineage-specific transcription factors, so that the disturbed expression or function of this group may be involved in the development of leukemia . PU.1 plays an important role in hematopiotic stem cell (HSC) self renewal and in myeloid and B-lymphoid differentiation. It controls the expression of several genes involved in hematopoiesis.

ELIGIBILITY:
Inclusion Criteria:

* children aged 2-17 years and diagnosed as new cases of acute lymphoblastic leukemia

Exclusion Criteria:

1. age more than 17 years
2. presence of other hematological disorders, history of other malignancies ,or relapsed ALL
3. patients under chemotherapy or radiotherapy

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * cases
    1. inclusion criteria: children aged 2-17 years and diagnosed as new cases of acute lymphoblastic leukemia
    2. exclusion criteria:
       1. age more than 17 years
       2. presence of other hematological disorders, history of other malignancies ,or relapsed ALL
       3. patients under chemotherapy or radiotherapy
  * controls (healthy age- and sex-matched children without ahistory of any malignancies)
Sampling Method: Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
FoxO3a and PU.1 levels in acute lymphoblastic leukemia | 2 years
  detection of the mean difference in FoxO3a and PU.1 expression levels between cases and controls

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferber EC, Peck B, Delpuech O, Bell GP, East P, Schulze A. FOXO3a regulates reactive oxygen metabolism by inhibiting mitochondrial gene expression. Cell Death Differ. 2012 Jun;19(6):968-79. doi: 10.1038/cdd.2011.179. Epub 2011 Dec 2. PMID 22139133
- [Background] Inaba H, Greaves M, Mullighan CG. Acute lymphoblastic leukaemia. Lancet. 2013 Jun 1;381(9881):1943-55. doi: 10.1016/S0140-6736(12)62187-4. Epub 2013 Mar 22. PMID 23523389
- [Background] Kerdiles YM, Beisner DR, Tinoco R, Dejean AS, Castrillon DH, DePinho RA, Hedrick SM. Foxo1 links homing and survival of naive T cells by regulating L-selectin, CCR7 and interleukin 7 receptor. Nat Immunol. 2009 Feb;10(2):176-84. doi: 10.1038/ni.1689. Epub 2009 Jan 11. PMID 19136962
- [Background] Pui CH. Acute lymphoblastic leukemia: introduction. Semin Hematol. 2009 Jan;46(1):1-2. doi: 10.1053/j.seminhematol.2008.09.011. No abstract available. PMID 19100362
- [Background] Xie Y, Davies SM, Xiang Y, Robison LL, Ross JA. Trends in leukemia incidence and survival in the United States (1973-1998). Cancer. 2003 May 1;97(9):2229-35. doi: 10.1002/cncr.11316. PMID 12712476
- [Background] Yang XB, Zhao JJ, Huang CY, Wang QJ, Pan K, Wang DD, Pan QZ, Jiang SS, Lv L, Gao X, Chen HW, Yao JY, Zhi M, Xia JC. Decreased expression of the FOXO3a gene is associated with poor prognosis in primary gastric adenocarcinoma patients. PLoS One. 2013 Oct 23;8(10):e78158. doi: 10.1371/journal.pone.0078158. eCollection 2013. PMID 24194912
- [Background] Zhang X, Tang N, Hadden TJ, Rishi AK. Akt, FoxO and regulation of apoptosis. Biochim Biophys Acta. 2011 Nov;1813(11):1978-86. doi: 10.1016/j.bbamcr.2011.03.010. Epub 2011 Mar 31. PMID 21440011
- [Result] Ausserlechner MJ, Salvador C, Deutschmann A, Bodner M, Viola G, Bortolozzi R, Basso G, Hagenbuchner J, Obexer P. Therapy-resistant acute lymphoblastic leukemia (ALL) cells inactivate FOXO3 to escape apoptosis induction by TRAIL and Noxa. Oncotarget. 2013 Jul;4(7):995-1007. doi: 10.18632/oncotarget.953. PMID 23828551
- [Result] Chiaretti S, Zini G, Bassan R. Diagnosis and subclassification of acute lymphoblastic leukemia. Mediterr J Hematol Infect Dis. 2014 Nov 1;6(1):e2014073. doi: 10.4084/MJHID.2014.073. eCollection 2014. PMID 25408859